CLINICAL TRIAL: NCT00307333
Title: Impact of Heart Rate Characteristics Monitoring in Neonates
Acronym: HeRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Medical Predictive Science Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10845
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Sepsis
Keywords: very low birth weight infants; heart rate characteristics
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Very low birth weight infants with their HRC index continuously displayed. Clinicians can utilize the HRC score to develop treatment plan.
  Interventions: Device: HeRO heart rate characteristics monitor
- 2 (No Intervention): Very low birth weight infants for whom the HRC index is not displayed. Infants receive standard of care treatment.

INTERVENTIONS:
Device: HeRO heart rate characteristics monitor — 24 hour continuous HRC monitoring with display
  Arms: 1

SUMMARY:
Hypothesis: Fewer neonates managed using information from heart rate characteristics (HRC) will require intubation and mechanical ventilation as a result of sepsis and sepsis-like illness.

Infants will be randomly assigned to one of two groups. One group of infants will have the HRC index known to the physicians caring for them, and physicians will use the HRC index as they desire to aid in clinical management.

Infants in the other group will have the HRC index recorded, but this information will not be displayed to the physicians caring for the infants.

DETAILED DESCRIPTION:
Following randomization, infants will be managed as usual practice. The treating physicians of the HRC-display group will be able to utilize the HRC score to assist in the care of the infant. The physicians of the no-display group will provide care as per standard.

Clinical symptoms will be treated according to the medical discretion of each physician. Cultures will be obtained and antibiotics administered as per the medical discretion of the physicians.

Clinical, culture results, antibiotic administration, ventilator use, and outcome at 120 days data will be collected on the infants as well as their HRC score calculated by the HeRO heart rate characteristics monitor.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to NICU
* Birth weight < 1500 grams
* Gestational age < or = 32 weeks
* Informed consent obtained from parent

Exclusion Criteria:

* Evidence of sustained cardiac arrhythmia
* Use of an electronic pacemaker

Ages: 1 Day to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3003 (Actual)
Dates: Start 2005-08; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Moorman, MD, Principal Investigator — University of Virginia
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Miami, Miami, Florida
  - Winnie Plamer Hospital for Women and Babies, Orlando, Florida
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] King WE, Carlo WA, O'Shea TM, Schelonka RL; HRC neurodevelopmental follow-up investigators. Multivariable Predictive Models of Death or Neurodevelopmental Impairment Among Extremely Low Birth Weight Infants Using Heart Rate Characteristics. J Pediatr. 2022 Mar;242:137-144.e4. doi: 10.1016/j.jpeds.2021.11.026. Epub 2021 Nov 17. PMID 34798080
- [Derived] King WE, Carlo WA, O'Shea TM, Schelonka RL; HRC neurodevelopmental follow-up investigators. Heart rate characteristics monitoring and reduction in mortality or neurodevelopmental impairment in extremely low birthweight infants with sepsis. Early Hum Dev. 2021 Aug;159:105419. doi: 10.1016/j.earlhumdev.2021.105419. Epub 2021 Jul 4. PMID 34247026
- [Derived] Swanson JR, King WE, Sinkin RA, Lake DE, Carlo WA, Schelonka RL, Porcelli PJ, Navarrete CT, Bancalari E, Aschner JL, Perez JA, O'Shea TM, Walker MW. Neonatal Intensive Care Unit Length of Stay Reduction by Heart Rate Characteristics Monitoring. J Pediatr. 2018 Jul;198:162-167. doi: 10.1016/j.jpeds.2018.02.045. Epub 2018 Apr 24. PMID 29703576
- [Derived] Sullivan BA, Grice SM, Lake DE, Moorman JR, Fairchild KD. Infection and other clinical correlates of abnormal heart rate characteristics in preterm infants. J Pediatr. 2014 Apr;164(4):775-80. doi: 10.1016/j.jpeds.2013.11.038. Epub 2014 Jan 10. PMID 24412138
- [Derived] Moorman JR, Carlo WA, Kattwinkel J, Schelonka RL, Porcelli PJ, Navarrete CT, Bancalari E, Aschner JL, Whit Walker M, Perez JA, Palmer C, Stukenborg GJ, Lake DE, Michael O'Shea T. Mortality reduction by heart rate characteristic monitoring in very low birth weight neonates: a randomized trial. J Pediatr. 2011 Dec;159(6):900-6.e1. doi: 10.1016/j.jpeds.2011.06.044. Epub 2011 Aug 24. PMID 21864846

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Very low birth weight infants with their HRC index continuously displayed. Clinicians can utilize the HRC score to develop treatment plan.
- Control: Very low birth weight infants for whom the HRC index is not displayed. Infants receive standard of care treatment.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 1511 | 1492
Completed | 1500 | 1489
Not Completed | 11 | 3
Not completed — Lost to Follow-up | 11 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 1511 | 1492 | 3003
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1511 | 1492 | 3003
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] — correct as reported
  years | 0.54 (0.054) | 0.54 (0.054) | 0.54 (0.054)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 791 | 767 | 1558
  Male | 720 | 725 | 1445
Region of Enrollment [Number; unit: participants]
  United States | 1511 | 1492 | 3003

OUTCOME MEASURES:

1. Primary Outcome: Number of Ventilator-free Days
Time Frame: 120 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1500 | 1489
days | 95.9 (35.1) | 93.6 (37.8)
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority or Other; p = 0.08, t-test, 2 sided

2. Secondary Outcome: Duration of Hospital Stay
Time Frame: 120 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1511 | 1492
days | 59.6 (33.7) | 58.7 (34.5)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority or Other; p = 0.47, t-test, 2 sided

3. Secondary Outcome: Days on Antibiotics
Time Frame: 120 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1500 | 1489
days | 15.7 (19.4) | 15.0 (19.1)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority or Other; p = 0.31, t-test, 2 sided

4. Secondary Outcome: Mortality
Time Frame: 120 days
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1500 | 1489
participants | 122 | 152
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority or Other; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.61 to 0.99] — HR = hazard for intervention / hazard for control

ADVERSE EVENTS:
Time Frame: 120 days follow-up
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 122/1500 | 152/1489
Other Adverse Events (participants affected / at risk) | 0/1500 | 0/1489
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=1500) | Control (N=1489)
Mortality [120 days] (Investigations) | 122 (122) | 152 (152)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No